CLINICAL TRIAL: NCT02861183
Title: A Randomized, Double-Blind, Placebo Controlled, Multi-Center Study of Sodium Hyaluronate to Provide Symptomatic Relief of Lateral Epicondylosis (Tennis Elbow)
Brief Title: Study of Sodium Hyaluronate to Provide Symptomatic Relief of Lateral Epicondylosis (Tennis Elbow)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project was placed on hold indefinitely as the project resources were unavailable for this to move forward.
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OVT 16-01
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Epicondylitis; Tennis Elbow; Epicondylosis
Keywords: sodium hyaluronate; OVT; hyaluronic acid
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- OVT (Sodium Hyaluronate) (Experimental): Sodium hyaluronate is supplied as a 2 mL unit dose in a 3 mL glass syringe.
  Interventions: Device: OVT (Sodium Hyaluronate)
- Saline (Placebo Comparator): 0.9% sterile saline is supplied as a 2 mL unit dose in a 3 mL glass syringe.
  Interventions: Device: Saline

INTERVENTIONS:
Device: OVT (Sodium Hyaluronate) — A Peri-osteotendinous injection of OVT will be administered into the soft tissue 1 cm from the lateral epicondyle at the point of greatest pain in two planes using a fanning technique. Two injections will be performed with a 22-25 gauge needle and spaced one week apart.
  Arms: OVT (Sodium Hyaluronate)
Device: Saline — A Peri-osteotendinous injection of sterile saline will be administered into the soft tissue 1 cm from the lateral epicondyle at the point of greatest pain in two planes using a fanning technique. Two injections will be performed with a 22-25 gauge needle and spaced one week apart.
  Arms: Saline

SUMMARY:
A Randomized, Double-Blind, Placebo Controlled, Multi-Center Study of Sodium Hyaluronate to provide Symptomatic Relief of Lateral Epicondylosis (Tennis Elbow).

DETAILED DESCRIPTION:
The objective of this study is to assess the safety and effectiveness of two weekly peri-osteotendinous injections of OVT for relief of pain in patients with lateral epicondylosis in a multi-center, randomized, double-blind, placebo controlled superiority study. A total of 186 subjects will be enrolled at up to 20 centers in the US and Europe. The randomization ratio will be 2:1 (2 OVT subjects: 1 placebo subject). The entire study duration from first subject in to last subject out is approximately one year. The enrollment phase is approximately 6 months with a follow-up phase of 6 months. Visits are scheduled at baseline, 1 week, 4 weeks, 12 weeks, 18 weeks, and 26 weeks. Study injections will be given at the baseline and 1 week visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 65 years of age
2. Clinical diagnosis of unilateral lateral epicondylosis defined as:

   1. Pain reproducible on palpation of the lateral epicondyle / common extensor origin; and
   2. Pain reproducible during resisted wrist extension
3. Subject is symptomatic for at least 6 weeks
4. Subject has pain in the index lateral epicondyle after grip strength testing that measures ≥ 40 mm on a 100 mm VAS
5. Subject must be willing to abstain from other pharmacological and surgical treatments of the index elbow for the duration of the study
6. Subject is willing to discontinue all systemic and/or topical analgesics including NSAIDs, (except the rescue medication oral acetaminophen/paracetamol), for the treatment of lateral epicondylosis at least seven days before the initial treatment injection and through the completion of the study
7. If pain medication is needed during the study, subject is willing to use only acetaminophen/paracetamol (up to a maximum of 3.0 grams per day per the package insert) for the treatment of elbow pain for the duration of the study
8. At least twenty four hours prior to the Baseline Visit and each follow-up visit, the subject must discontinue use of acetaminophen/paracetamol, if used
9. Subject is able to understand and comply with the requirements of the study and voluntarily provides consent

Exclusion Criteria:

1. Subjects with a history of hypersensitivity to any of the ingredients in the hyaluronan or an inability to tolerate acetaminophen/paracetamol
2. Subjects in which the investigator believes the anatomical landmarks for injection are unable to be adequately identified
3. Subjects who have a history of surgery to the intra-articular joint of the index elbow and/or history of index elbow dislocation
4. Any diagnosed pathology or trauma that causes pain or symptoms in the index elbow other than lateral epicondylosis (e.g. intra-articular pathology, ligament injury, cervical radiculopathy, radial tunnel syndrome, osteochondral radiocapitellar lesion or posterolateral elbow plica, pain starting after a motor vehicle accident)
5. Hyaluronic acid injections in the index elbow within the last 6 months
6. Steroid injections in the index elbow within the last 3 months
7. Infections or skin diseases in the area of the injection site or elbow joint
8. Known inflammatory or autoimmune disorders, or other pre-existing medical conditions that, in the opinion of the investigator, could impact healing or affect the ability of the subject to complete the study and comply with the study requirements
9. Subject is taking medications at the time of consent which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment and opioid analgesics. Low dose aspirin (81 mg) used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
10. Subject is receiving or in litigation for worker's compensation
11. Subject is a woman who is pregnant or breastfeeding at the screening visit or a woman of child bearing potential who refuses to use effective contraception during the course of the study
12. Subject was involved in any other research study involving an investigational product, or a new application of an approved product, within 60 days of signing the Informed Consent Form (ICF)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in elbow pain after grip as measured by a 100 mm Visual Analog Scale (VAS) at 12 weeks comparing the OVT group to the saline control group | 12 weeks post injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.

SECONDARY OUTCOMES:
The change from baseline in elbow pain after grip as measured by a 100 mm VAS at 4, 18, and 26 weeks comparing the OVT group to the saline control group | 4, 18, 26 weeks post-injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.
The change from baseline in elbow pain after grip as measured by a 100 mm VAS through 4-26 weeks using a longitudinal model comparing the OVT group to the saline control group | 26 weeks post-injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.
The change from baseline in elbow pain at rest as measured by a 100 mm VAS through 4-26 weeks using a longitudinal model comparing the OVT group to the saline control group | 26 weeks post-injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.
The change from baseline in elbow pain as measured by the Patient-Rated Tennis Elbow Evaluation (PRTEE) Pain and Function Questionnaire through 4-26 weeks using a longitudinal model comparing the OVT group to the saline control group | 26 weeks post-injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.
The change from baseline in elbow pain as measured by the Disabilities of Arm, Shoulder, and Hand (DASH) Questionnaire through 4-26 weeks using a longitudinal model comparing the OVT group to the saline control group | 26 weeks post-injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.
The change from baseline in Grip Strength using a hydraulic hand dynamometer at 4, 12, 18, and 26 weeks comparing the OVT group to the saline control group | 4,12,18 and 26 weeks post-injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.
The change from baseline in rescue medication consumption (acetaminophen/ paracetamol) through weeks 4-26 comparing the OVT group to the saline control group | 26 weeks post-injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.
The incidence, timing, severity, and relationship to treatment of all adverse events will be classified using MedDRA. | During injection, 4, 12, 18 and 26 weeks post-injection
  Pain After Grip score was determined by asking the subject "How much pain do you have in your STUDY elbow right now?" and recording their response by placing a mark along a 100mm VAS scale with 0mm=no pain and 100mm=extreme pain. A negative value for change from baseline indicated a reduction in pain. A greater negative value indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: TBD TBD, Principal Investigator

IPD SHARING:
Plan to Share IPD: No